CLINICAL TRIAL: NCT03077152
Title: Patient Factors Associated With Prescription of Antibiotics for Inappropriate Indication in Patients With AECOPD
Status: Completed | Type: Observational
Sponsor: Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yelda Varol, Principal Investigator MD, Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital
Other Study IDs: IGHCEAH
Record Dates: First submitted 2017-02-28; First posted 2017-03-10 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Acute Exacerbation of COPD
Keywords: copd, aecopd, antibiotic use
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Up to 90% of consulting Acute Exacerbation (AE) of COPD patients are prescribed an antibiotic(1).

Rates of inappropriate antibiotic prescription percentage can be as high as 65%(2).

Excessive use of antibiotics is correlated with higher prevalence of antimicrobial resistance(3). There are insufficient data regarding the overprescribing antibiotics in AECOPD in our country.Therefore the investigators aimed to investigate the patients factors that are associated with the prescription of antibiotic for inappropriate indication in AECOPD.This is an observational cross sectional study.Population: AECOPD patients with AB(antibiotic) prescription Exposure: Presence of patient factors, Comparison: Absence of Patient factors, Outcome: Prescription of antibiotic for inappropriate indication.

Sampling:

Consecutive patients presenting to pharmacy between Monday and Friday. Date between January 1 2017 to January 1 30 2019. Primary Outcome:Prescription of antibiotic for inappropriate indication according to Anthonisen criteria for AECOPD Anthonisen criteria:-Worsening of dyspnea

* Increased sputum volume
* Increased sputum purulent 3/3 →Type 1 or severe AE 2/3 →Type 2 or moderate AE 1/3 →Type 3 or mild AE AB indicated/useful in Type 1 or severe AE, and Type 2 or moderate AE if sputum is purulent The data will be obtained from the database.

Exposure:

Patient factors that lead to inappropriate antibiotic prescription (will be considered together in analysis due to confounding) FEV1% Age Current smoker Comorbidities (Charlson comorbidity index) having Frequent exacerbations (≥2 past year) Use of oral steroids Polypharmacy Quality control:Detailed MOP will be developed, A manual for protocol will be written and used to inform the pharmacist,Pharmacist will be trained; to speak to participants in a neutral manner for written informed consent for the security ID(identity) data of the patients,This study will not affect the time period of the participants to access his/her drug. The pharmacy will use the questionnaire within the time period planned. A checklist for exclusion criteria will be developed. A plan for missing data will be developed.

Null hypothesis:

Patient factors are not associated with the prescription of antibiotics for inappropriate indications in patients with AECOPD

Alternative hypothesis:

Patient factors are associated with the prescription of antibiotics for inappropriate indications in patients with AECOPD Analysis The data will be analysed using SPSS version 22.0 The investigators will compare exposure variables between inappropriate and appropriate prescription groups Continuous variables - t test or Mann Whitney Binary- chi square test The investigators will use logistic regression to measure the associations between patient factors and the outcome of prescription of antibiotics for inappropriate indication Sample size and power Sample size to estimate CI of 15% around 25 to 50% prevalence of inappropriate prescription with p=0.05 and Power 80% Expected proportion0,25 128 0,50 171 Sample size and power For logistic regression - estimate 30% prevalence (n=143), or about 42 events . The investigators also need 5-10 events for each variable in the model, so this provides sufficient power for 4 to 8 factors.

Limitations This study will just determine an association not causality

The investigators won't be able to determine if the participant is truthful to the pharmacist

The history of participants will be assessed from hospitals e-database - potential for missing data.

The Anthonisen criteria for identifying inappropriate AB for AECOPD are still debatable The investigators can not modify many of the patient factors, but may be able to identify patients at higher risk of inappropriate antibiotics Ethics The project will be submitted to the ethical committee of Dr. Suat Seren Chest Disease Hospital Oral and written informed consent will be obtained from all subjects The study will be conducted in accordance with "Good Clinical Practice Guideline" Relevance This study will be the first one to evaluate an association between patient factors and prescription of antibiotic for inappropriate indication in an outpatient clinic of patients with AECOPD in Turkey.

Subsequent studies should evaluate physician factors prescription of antibiotic for inappropriate indication.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with COPD according to GOLD criteria
* Patients whom are prescripted an antibiotic for AECOPD in a chest diseases outpatient clinic
* Prescriptions should be written by pulmonologists

Exclusion Criteria:

* COPD patients using Long term oxygen treatment (LTOT) at home
* COPD patients using Bilevel Positive airway pressure (BPAP) for type 2 respiratory failure
* COPD patients whom have snother need for AB use (bronchiectasis Pneumonia etc.)
* COPD patients with Positive sputum culture past 4 weeks
* COPD patients whom have Hospitalisation for COPD past 4 weeks

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AECOPD patients with Antibiotic prescription
Sampling Method: Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Number of participants who has a prescription of antibiotic for inappropriate indication for AECOPD according to Anthonisen criteria | 3 months
  Prescription of antibiotic is indicated in type 1 or severe exacerbation (3/3 Antjonisen critaria) or type 2 or moderate exacerbation if one of the symptoms are purulens of sputum.In mild exacerbation (1/3 criteria) it is not indicated.

SECONDARY OUTCOMES:
Patient factors that may lead to prescribe inappropriate antibiotic prescription | 6 months
  Probable Patient factors that lead to inappropriate antibiotic prescription are FEV1%, Age, being a current smoker, carlson comorbidity index, being a frequent exacerbator, use of oral steroids and polifarmacy (will be considered together in analysis due to confounding)

CONTACTS AND LOCATIONS:
Overall Officials: Yelda Varol, MD, Principal Investigator — Izmir Dr. Suat Seren Chest Diseases and Surgery Education and Training Hospital
Locations (1):
- Dr. Suat Seren Chest Diseases and Surgery Education and Training Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Llor C, Bjerrum L, Munck A, Hansen MP, Cordoba GC, Strandberg EL, Ovhed I, Radzeviciene R, Cots JM, Reutskiy A, Caballero L. Predictors for antibiotic prescribing in patients with exacerbations of COPD in general practice. Ther Adv Respir Dis. 2013 Jun;7(3):131-7. doi: 10.1177/1753465812472387. Epub 2013 Jan 16. PMID 23325784
- [Background] Tobia CC, Aspinall SL, Good CB, Fine MJ, Hanlon JT. Appropriateness of antibiotic prescribing in veterans with community-acquired pneumonia, sinusitis, or acute exacerbations of chronic bronchitis: a cross-sectional study. Clin Ther. 2008 Jun;30(6):1135-44. doi: 10.1016/j.clinthera.2008.06.009. PMID 18640469
- [Background] Bronzwaer SL, Cars O, Buchholz U, Molstad S, Goettsch W, Veldhuijzen IK, Kool JL, Sprenger MJ, Degener JE; European Antimicrobial Resistance Surveillance System. A European study on the relationship between antimicrobial use and antimicrobial resistance. Emerg Infect Dis. 2002 Mar;8(3):278-82. doi: 10.3201/eid0803.010192. PMID 11927025
- [Background] Anthonisen NR, Manfreda J, Warren CP, Hershfield ES, Harding GK, Nelson NA. Antibiotic therapy in exacerbations of chronic obstructive pulmonary disease. Ann Intern Med. 1987 Feb;106(2):196-204. doi: 10.7326/0003-4819-106-2-196. PMID 3492164